CLINICAL TRIAL: NCT06191718
Title: Clinical Investigation for the Foldax Tria Mitral Valve- India
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foldax, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-004
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Mitral Valve Disease; Mitral Regurgitation; Mitral Stenosis; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tria Mitral Valve (Experimental): Patients receiving the Foldax Mitral Valve
  Interventions: Device: Mitral Valve Replacement

INTERVENTIONS:
Device: Mitral Valve Replacement — Foldax Mitral Valve Replacement

SUMMARY:
The purpose of this study is to conduct a clinical investigation of the Foldax Tria Mitral Valve to collect evidence on the device's safety and performance.

DETAILED DESCRIPTION:
The Foldax Tria Mitral Heart Valve is indicated as a replacement for diseased, damaged, or malfunctioning native mitral heart valve via open heart surgery. The study is a single open are label non-randomized multi- center clinical trial. Up to 10 sites in the country of India will enroll up to 70 patients. The first two patients at each site, will be considered roll-in patients accounting for training. Up to 50 patients will be considered part of the treatment phase. These patients will follow the study schedule for 1 year after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older
* Is a candidate for mitral valve replacement with cardiopulmonary bypass
* Is a candidate for mitral valve replacement due to severe mitral valve disease
* No contraindication for anticoagulation treatment
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Requires valve replacement other than mitral
* Prior mitral valve surgery for valve replacement or valve repair (this does NOT include percutaneous interventions i.e. Mitraclip, chordal replacement)
* Required concomitant cardiovascular procedures except for CABG and/or COX-MAZE if approved by the screening committee
* Requires emergency surgery
* Requires other planned surgery within 12 months of valve replacement
* Active endocarditis or active myocarditis
* Exhibits left ventricular ejection fraction </= 20% as validated by diagnostic procedure prior to planned valve surgery
* Acute preoperative neurological deficit defined as neurological deficit < 3 months prior to enrollment
* Life expectancy of less than 12 months
* Enrolled in another investigational device or drug study (enrolled patients may not enroll in other studies)
* Myocardial infarction, or severe cardiac adverse event which has not returned to baseline for at least 30-days prior to enrollment
* Aortic aneurysm or other medical condition that creates a higher than usual risk of surgical complications
* Renal insufficiency as determined by creatinine (S-CR) level as >/= 2.0 mg/dl or end stage renal disease requiring chronic dialysis at screening visit
* Results for the following blood tests are not within normal limits: D-Dimer, Basic Metabolic Panel Liver enzymes, Coagulation Profile - platelets, APTT, INR, Fibrinogen, C-reactive protein (HSCRP) and ESR, and Troponin levels
* Hematological disorders, patients must not have a hematocrit of <30%, hemoglobin <10 g/dL, platelet count of <100,000 cells/µL, or WBC <4,000 cells/µL; coagulation profile must not be outside of normal limits
* Patients who are pregnant or expect to become pregnant in the 12 months following implantation, or are lactating
* Any other condition that, in the judgment of the investigator and screening committee, makes the patient a poor candidate for the procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, extensive travel away from the research center, COVID-19 related concerns)
* Patients who have withdrawn after implantation may not re-enter
* Intraoperatively it is determined that the patient anatomy is not compatible with the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints | 12 months after last patient enrollment
  Serious Adverse Event (SAE) rates for any valve related events. Results are compared descriptively to event rates reported in the literature.
Primary Effectiveness Endpoint- Change in Hemodynamic Performance | 12 months after last patient enrollment
  Hemodynamic performance parameters are mmHG mean gradient, peak gradient, and derived Effective Orifice Area (EOA). Success is defined as clinically significant improvement in hemodynamic performance (mean/peak gradient and Effective Orifice Area (EOA)) at one year based on literature reports for surgical mitral valve replacement.
Clinical Effectiveness Endpoint- Change in New York Heart Association Assessment | 12 months after last patient enrollment
  Clinically significant improvement (one grade) in the New York Heart Association (NYHA) functional classification status at 365 days compared to baseline. a. Class I - No symptoms and no limitations in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. b. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. c. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest. d. Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

SECONDARY OUTCOMES:
Number of Participants with Stroke | 1 year following patient enrollment
  Assessment of patient experiencing a stroke (ex; ischemic stroke, intracerebral hemorrhage, subarachnoid hemorrhage, or other) verified by imaging and or physical exam
Number of Participants with Structural Valve Deterioration (SVD) | 1 year following patient enrollment
  Assessment of patient experiencing SVD as verified by imaging, procedure, or physical exam
Number of Participants with Transient Ischemic Attack | 1 year following patient enrollment
  Assessment of patient having a TIA as verified by imaging and or physical exam
ICU Duration of Stay | 30 Days post patient enrollment
  Length of stay in the ICU post valve implantation defined as arrival time/date in hours and minutes to transfer to floor time/date in hours and minutes.
Ventilation Time | 30 Days post patient enrollment
  Ventilation time in hours defined as arrival time/date in recovery in hours and minutes to date and time extubated in hours and minutes
Post Procedure length of stay | 30 days post patient enrollment
  Post procedure length of stay defined as the time/date documented for arrival in the recovery unit to date/ time of discharge in hours and minutes.
Kansas City Cardiomyopathy Questionnaire | 12 months post patient enrollment
  Change in QOL as measured by the KCCQ. Scores are measured from 0-100, in hich higher scores reflect better health status.
Six Minute Walk Test | 12 months post patient enrollment
  Change in patients activity tolerance as documented by a 6 Minute Walk Test assessed by distance traveled after 6 minutes

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - GCS Medical College, Ahmedabad, Gujarat
  - Epic Hospital, Ahmedabad, Gujarat
  - KEM Hospital, Mumbai, Maharashtra
  - Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Six Sigma, Nashik, Maharashtra
  - B.J. Medical College, Pune, Maharashtra
  - SMS Hospital, Jaipur, Rajasthan
  - Indo-US Hospital, Hyderabad, Telangana
  - NRS Medical College and Hospital, Kolkata, West Bengal
  - Fortis Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] George I, Rao DP, Jain A, Ascione G, Sharma M, Meharwal ZS, Sarkar B, Kochar N, Gan MD, Shastri N, Runt J, Whisenant B, Wilson B, Kiser A, Leon MB, Pandey K. 1-Year Results From a Multicenter Trial of a Polymer Surgical Mitral Valve: Insights Into New Technology. J Am Coll Cardiol. 2025 Aug 19;86(7):515-526. doi: 10.1016/j.jacc.2025.06.017. Epub 2025 Jun 27. PMID 40589299